CLINICAL TRIAL: NCT03184246
Title: The Depth of Endotracheal Tube Insertion - Use of Direct Laryngoscopy and Videolaryngoscopy (GlideScope), Comparison of Methods
Brief Title: The Depth of Endotracheal Tube Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, MD, Ph.D., University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: University Hospital
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Intubation Complication
Keywords: Videolaryngoscopy (GlideScope); Direct laryngoscopy

STUDY DESIGN:
Intervention Model Description: Interventional group will be intubated by videolaryngoscopy, control group by direct laryngoscopy
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlideScope (Experimental): intubation with GlideScope
  Interventions: Device: GlideScope
- Direct laryngoscopy (Active Comparator): intubation with laryngoscope
  Interventions: Device: Direct laryngoscopy

INTERVENTIONS:
Device: GlideScope — videolaryngoscopy (GlideScope) will be used for intubation
  Arms: GlideScope
Device: Direct laryngoscopy — direct laryngoscopy will be used for intubation
  Arms: Direct laryngoscopy

SUMMARY:
The investigators suppose that direct laryngoscopy is connected with deeper insertion of endotracheal tube in comparison to videolaryngoscopy. Correction of this malposition can cause postoperative discomfort and further complications in some patients.Routine use of videolaryngoscopy could minimize these problems.

DETAILED DESCRIPTION:
100 patients scheduled for elective neurosurgical procedures will be randomized into two groups. Patients in group A will be intubated by videolaryngoscopy (GlideScope), patients in group B by direct laryngoscopy, in both groups will be rigid stylet used. Intubation will be done under propofol anesthesia, targeted entropy 40 to 50, and deep relaxation (neuromuscular transmission target level 0). Sufentanil will be used to block tracheal reflexes. In both groups the depth of insertion of tracheal tube will be measured in the mouth corner immediately after intubation. Next day, the unpleasant sensations and complications will be recorded (sore throat, stridor, hoarseness, cough and nausea and vomiting) during control visit of patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I - III

Exclusion Criteria:

* postoperative ventilation, laryngeal tumors, conditions after tracheotomy or laryngeal operations, cervical spinal hernia extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
the depth of primary insertion of tracheal tube | in a minute after intubation
  cm

SECONDARY OUTCOMES:
sums of manipulation with tracheal tube | 2 minutes after intubation
  number
complications after intubation | 24 hours after surgery
  number

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Dostal, MD, Ph.D., Study Director — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No